CLINICAL TRIAL: NCT00310167
Title: A Phase III Multi-Center Randomized Controlled Trial of Low-Dose Radiotherapy for Follicular Lymphoma and Marginal Zone Lymphoma
Brief Title: Low-Dose Radiation Therapy in Treating Patients With Follicular or Marginal Zone Non-Hodgkin's Lymphoma
Acronym: FoRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/05/84; CRUK-FORT; CRUK-BRD/05/84; 2005-002416-19 (EudraCT Number); ISRCTN65687030; EU-20601
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; Marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4 Gy (Experimental): 4 Gy in 2 fractions
  Interventions: Radiation: radiation therapy
- 24 Gy (Active Comparator): 24 Gy in 12 fractions
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill cancer cells. It is not yet known which regimen of low-dose radiation therapy is more effective in treating follicular non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two different regimens of low-dose radiation therapy (24Gy versus 4Gy) to compare how well they work in treating patients with follicular or marginal zone non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the local progression-free interval in patients with follicular non-Hodgkin's lymphoma (NHL) treated with 2 different regimens of low-dose radiotherapy.

Secondary

* Compare acute toxicity at 4 weeks in patients treated with these regimens.
* Compare late toxicity in patients treated with these regimens.
* Compare tumor response at 12 weeks in patients treated with these regimens.
* Compare overall survival in patients treated with these regimens.
* Assess the health economics of these regimens in these patients.

OUTLINE: This is a multicenter, randomized study. Patients are randomized to one of two treatment arms.

* Arm I 4Gy: Patients undergo low-dose radiotherapy once daily on days 1 and 2.
* Arm II 24Gy: Patients undergo low-dose radiotherapy once daily on days 1-5, 8-12, 15, and 16.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 650 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed follicular or mmarginal zone non-Hodgkin's lymphoma (NHL)

  * Any stage
* Radiotherapy is indicated for curative treatment of stage IA or IIA disease OR palliation due to tumor bulk or anatomical position

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2005-10; Primary Completion 2013-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Local progression-free interval in irradiated field | up to 5 years after randomisation
  Time form randomisation to tumour progression within the irradiated field

SECONDARY OUTCOMES:
Acute toxicity | at 4 weeks after randomization
Late toxicity | from 12 weeks after randomisation up to 5 years
Tumor response in irradiated area at 12 weeks after randomization | at 12 weeks after randomization
Overall survival | up to 5 years after randomisation
Health economic assessment | up to 5 years after randomisation

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Research UK and University College London Cancer Trials Centre, London, England, United Kingdom

REFERENCES:
- [Derived] Hoskin P, Popova B, Schofield O, Brammer C, Robinson M, Brunt AM, Madhavan K, Illidge T, Gallop-Evans E, Syndikus I, Clifton-Hadley L, Kirkwood AA. 4 Gy versus 24 Gy radiotherapy for follicular and marginal zone lymphoma (FoRT): long-term follow-up of a multicentre, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2021 Mar;22(3):332-340. doi: 10.1016/S1470-2045(20)30686-0. Epub 2021 Feb 1. PMID 33539729
- [Derived] Hoskin PJ, Kirkwood AA, Popova B, Smith P, Robinson M, Gallop-Evans E, Coltart S, Illidge T, Madhavan K, Brammer C, Diez P, Jack A, Syndikus I. 4 Gy versus 24 Gy radiotherapy for patients with indolent lymphoma (FORT): a randomised phase 3 non-inferiority trial. Lancet Oncol. 2014 Apr;15(4):457-63. doi: 10.1016/S1470-2045(14)70036-1. Epub 2014 Feb 24. PMID 24572077